CLINICAL TRIAL: NCT05451212
Title: A Phase 1, Open-label, Safety and Dose-finding Study of Autologous Muscle-specific Tyrosine Kinase Chimeric Autoantibody Receptor T Cells (MuSK-CAART) in Subjects With Anti-MuSK-antibody-positive Myasthenia Gravis
Brief Title: Open-label Study to Evaluate the Safety of Various Dosing Regimens of MuSK-CAART for MuSK Myasthenia Gravis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cabaletta Bio (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAB-MuSK-101
Record Dates: First submitted 2022-06-30; First posted 2022-07-11 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: MuSK Myasthenia Gravis
Keywords: CAAR-T (Chimeric Autoantibody Receptor T Cells) Therapy; CAR-T (Chimeric Antigen Receptor T Cells) Therapy; Cell Therapy; Autoimmune Disease; Autoimmunity; Immunotherapy, Adoptive; Immune System Diseases; Myasthenia Gravis (MG); Muscle-specific tyrosine kinase (MuSK); Muscle Weakness; Neuromuscular Diseases; Musculoskeletal Diseases
MeSH Terms: conditions — Myasthenia Gravis; Autoimmune Diseases; Immune System Diseases; Muscle Weakness; Neuromuscular Diseases; Musculoskeletal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MuSK-CAART (Experimental): Cohort A: Infusion of MuSK-CAART at various dose levels with or without pre-treatment (6 groups planned).
  Cohort B: Infusion of MuSK-CAART at the dose regimen selected from Part A.
  Interventions: Biological: MuSK-CAART

INTERVENTIONS:
Biological: MuSK-CAART — Intravenous infusion of MuSK-CAART at different doses. Subjects may also receive MuSK-CAART following pre-treatment with CY, or CY plus FLU.

SUMMARY:
Muscle-specific tyrosine kinase (MuSK) myasthenia gravis (MG) is a rare but potentially severe disease, in which patients develop pathogenic autoantibodies that specifically target the MuSK protein in the neuromuscular junction. This phase 1 study is being conducted to evaluate the safety of various dosing regimens of an investigational cell therapy, MuSK-CAART, that can be given to patients with anti-MuSK antibody positive Myasthenia Gravis (MuSK MG), who have active disease. Various dosing regimens of MuSK-CAART alone, in combination with cyclophosphamide (CY), and in combination with CY and fludarabine (FLU) will be evaluated. Treatment with MuSK-CAART may potentially lead to complete and durable remission of disease.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of MuSK-type MG with at least 1 prior positive anti-MuSK antibody test.
* History of a negative anti-AChR (acetylcholine receptor) antibody test.
* Positive anti-MuSK antibody test at screening
* MG severity Class I to IVa on the MGFA (Myasthenia Gravis Foundation of America) Clinical Classification

Exclusion Criteria:

* Rituximab in the last 12 months.
* Prednisone > 0.25mg/kg/day [in Part A]
* Other autoimmune disorder requiring immunosuppressive therapies.
* Investigational treatment for MG in the past 12 weeks.
* Absolute lymphocyte count < 500/µL at screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2022-11-23 (Actual); Primary Completion 2025-07-24 (Actual); Study Completion 2025-07-24 (Actual)

PRIMARY OUTCOMES:
Adverse events | 3 months
  Incidence of adverse events (AEs), including dose-limiting toxicities (DLTs) and AEs that are related to MuSK-CAART.

SECONDARY OUTCOMES:
Total MuSK-CAART positive cells | Baseline
  Total MuSK-CAART positive cells for each manufacturing run.
Percent of CAAR-transduced cells | Baseline
  Percent of total cells for infusion that are CAAR (Chimeric Autoantibody Receptor)-transduced cells.
Cellular kinetics profile of MuSK-CAART | Up to 36 months
  Cellular kinetics profile of MuSK-CAART after infusion.
Change in MuSK autoantibody titer | Up to 36 months
  Change in MuSK autoantibody titer compared to pre-infusion visit by clinically validated assay.

OTHER OUTCOMES:
Use of Concomitant Therapies | Up to 36 months
  Frequency and dose of concomitant therapies.
Measurement of Clinical Symptoms using MG-ADL | Up to 36 months
  Measurement of clinical symptoms using the Myasthenia Gravis Activities of Daily Living (MG-ADL) assessment.
Measurement of Clinical Symptoms using QMG | Up to 36 months
  Measurement of clinical symptoms using the Quantitative Myasthenia Gravis (QMG) assessment.
Measurement of Clinical Symptoms using MGC | Up to 36 months
  Measurement of clinical symptoms using the Myasthenia Gravis Composite (MGC) assessment.
Measurement of Quality of Life (QoL) using MG-QOL-15r | Up to 36 months
  Measurement of Quality of Life using the MG-QOL-15r (Myasthenia Gravis Qualify of Life 15-item scale, revised) questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Chair — Cabaletta Bio
Locations (5):
- United States (5):
  - UC Irvine, Department of Neurology, Orange, California
  - UC Davis, Department of Neurology, Sacramento, California
  - University of Kansas Medical Center, Kansas City, Kansas
  - Oregon Health & Science University (OHSU), Portland, Oregon
  - Houston Methodist Hospital, Houston, Texas